CLINICAL TRIAL: NCT03930966
Title: Study of the Association Between a Peri-traumatic Dissociation State and the Occurrence of Post-traumatic Stress Syndrome After Severe Trauma Requiring General Anesthesia
Brief Title: Association Between a Peri-traumatic Dissociation State and the Occurrence of Post-traumatic Stress Syndrome
Acronym: DIStress-AG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DIStress-AG (29BRC18.0200)
Record Dates: First submitted 2019-02-28; First posted 2019-04-29 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-09

CONDITIONS: Severe Trauma; General Anaesthesia
Keywords: Severe trauma; General anaesthesia; Peri-traumatic dissociation state; Post-traumatic stress disorder
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Prospective Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDEQ, PCL-5 and demographic survey (Experimental): State of the patient evaluated with questionnaires to make the connection between peri-traumatic dissociation and the occurrence of post-traumatic stress disorder
  Interventions: Diagnostic Test: PDEQ, PCL-5 and demographic survey

INTERVENTIONS:
Diagnostic Test: PDEQ, PCL-5 and demographic survey — Questionnaires

SUMMARY:
Patients will be selected after studying clinical records.Patients who had general anesthesia due to an injury related to severe trauma within 6 to 12 months prior to inclusion will be included.

Three self-survey will be completed by the patient: PDEQ, PCL-5 and a demographic questionnaire. According to the PDEQ and PCL-5 scores, an association between a peri-traumatic dissociation state and a post-traumatic stress disorder can be established.

ELIGIBILITY:
Inclusion Criteria:

* Patients with general anesthesia for a surgical wound with violent trauma in the road, a fall of more than 6 meters, burn, accident at work, explosion, aggression) in the 6 to 12 months before the inclusion
* Time between trauma and general anesthesia should not exceed 48 hours
* Patient agreeing to participate in the study.

Exclusion Criteria:

* Minor patients
* Patients under curatorship, and tutorship
* Patient deprived of liberty
* Patients who do not speak French
* Patients who are not in satisfactory neurological state to answer the questionnaire (pyschotic, demented states)
* Patients who have been sedated (apart from general anesthesia) when receiving or having a Glasgow score <14

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Studying association between the presence of peri-traumatic dissociation state and the achievement of post-traumatic stress disorder between 6 and 12 months in traumatized patients | study baseline (6 to 12 months after initial hospitalisation)
  Association will be measured using PDEQ scale and PCL-5 scale. The peri-traumatic dissociation will be evaluated by the Peri-traumatique Dissociation Experience Questionnary (PDEQ scale). This questionnaire contains ten items to study the presence or not of a peri-traumatic dissociation state. The items are scored on a 5-point Likert scale ranging from 1 (not at all true) to 5 (extremely true). The total score is the sum of all the items. A score from 15 indicates a significant dissociation.
  The presence or not of a Post-Traumatic Stress Disorder (PTSD) will be evaluated by the Post-Traumatic Stress Disorder Checklist Scale-Version DSM 5 (PCL-5). This questionnaire contains twenty items to study the presence or not of a PTSD. A total score for symptom severity (0-80) can be obtained by summing the scores for each of the 20 items. A score over 31 indicates a PTSD.

SECONDARY OUTCOMES:
Measurement of the frequency of PTSD after severe trauma requiring general anesthesia. | study baseline (6 to 12 months after initial hospitalisation)
Research of Risk Factors Associated with the Occurrence of PTSD | study baseline (6 to 12 months after initial hospitalisation)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ARIES, Dr, Principal Investigator — philippe.aries@chu-brest.fr
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.